CLINICAL TRIAL: NCT05338788
Title: Balance Performance in Dual Task in Patients With Cervical Disc Herniation Related Chronic Neck Pain: a Comparative Study
Brief Title: Balance Performance in Dual Task in Patients With Cervical Disc Herniation Related Chronic Neck Pain:a Comparative Study
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IzmirBozyaka-HayriyeYILMAZ-001
Record Dates: First submitted 2022-04-05; First posted 2022-04-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cervical Pain; Postural Balance
Keywords: Cervical Pain; postural balance; Biodex Balance System; Cervical disc herniation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Thirty-two 32 patients with cervical disk herniation related chronic neck pain participated in this cross-sectional controlled study. Patients who aged 18-64 years, had neck pain for at least 12 weeks, no tumor, trauma, fracture pathology in the spinal region and no history of spine surgery were included.
  The Neck Disability Index (NDI) was used to assess neck pain related disability. The Biodex Balance System (BBS; Biodex Medical Systems, Shirley, New York, USA) was used to assess postural control. The evaluated parameters of this system are presented below: modified clinical test of sensory integration of balance (mCTSIB), athletic single leg test (ASLT), limits of stability (LOS), and fall risk assessment were performed with and without a cognitive task. Dual-task interference (DTI) was assessed.
  Interventions: Other: neck pain and dual task
- Control Group: Twenty-three 23 age and sex-matched asymptomatic controls participated in this cross-sectional controlled study.
  The Biodex Balance System (BBS; Biodex Medical Systems, Shirley, New York, USA) was used to assess postural control.The evaluated parameters of this system are presented below: modified clinical test of sensory integration of balance (mCTSIB), athletic single leg test (ASLT), limits of stability (LOS), and fall risk assessment were performed with and without a cognitive task. Dual-task interference (DTI)was assessed.
  Interventions: Other: neck pain and dual task

INTERVENTIONS:
Other: neck pain and dual task — The Neck Disability Index (NDI) was used to assess neck pain related disability. The Biodex Balance System was used to assess postural control.Clinical test of sensory integration of balance (mCTSIB), athletic single leg test (ASLT), limits of stability (LOS), and fall risk assessment were performed with and without a cognitive task.In order to avoid the order bias of postural control measurements during "Single-task" and "Dual-task" for each case, the order of the measurements was determined by randomization on the first day by using sealed envelope method. After single/double task randomization was made, the order of tests was also randomized by using sealed envelopes containing two different orders (1-mCTSIB, 2-ASLT, 3-Fall test, 4-LOS and 1- LOS, 2- Fall test, 3- ASLT, 4-mCTSIB).

SUMMARY:
Intense pain and moderate disability are seen most patients with symptomatic cervical disc herniation (CDH). Since neck motion and motor control are associated with changes in neck pain and disability, it is highly likely that patients with neck pain related disability would display dual-task interference (DTI) during postural control with a cognitive task.

It is very important for patients with cervical disk herniation to perform more than one task at the same time for many activities of daily living. Therefore, the aim of this study was to compare balance performance in dual task between patients with CDH related chronic neck pain and asymptomatic controls.

DETAILED DESCRIPTION:
This study was designed cross-sectional controlled study. Thirty-two patients with CDH related chronic neck pain and twenty-three age and sex-matched asymptomatic controls participated in this study.

The Neck Disability Index (NDI) was used to assess neck pain related disability. The Biodex Balance System (BBS; Biodex Medical Systems, Shirley, New York, USA) was used to assess postural control. This system allows individuals to measure their stability limits. It also examines the control of the center of gravity on the support surface and balance abilities when trying to move it. The evaluated parameters of this system are presented below; modified clinical test of sensory integration of balance (mCTSIB), athletic single leg test (ASLT), limits of stability (LOS), and fall risk assessment were performed with and without a cognitive task. Dual-task interference (DTI) was assessed.

In order to avoid the order bias of postural control measurements during "Single-task" and "Dual-task" for each case, the order of the measurements was determined by randomization on the first day by using sealed envelope method. After single/double task randomization was made, the order of tests was also randomized by using sealed envelopes containing two different orders (1-mCTSIB, 2-ASLT, 3-Fall test, 4-LOS and 1- LOS, 2- Fall test, 3- ASLT, 4-mCTSIB).

Before starting the evaluations, the participants were informed about the tests. Considering methodological bias, the same investigator performed all assessments and all participants received standardized and identical instructions.

Single and dual task measurements were made as follows:

Single task measurements involved the measurement of balance parameters by using Biodex Balance System without any additional cognitive task. For assessment of dual task performance, the participants were asked to perform an additional cognitive task (counting backwards from 200 by three or seven) during measurements .

DTI values were calculated for all balance parameters using the formulas below :

DTI %= (Dual Task-Single Task)/Single Task*100

ELIGIBILITY:
Inclusion Criteria:

1.18 to 64 years of age 2.Having generalized neck pain for more than 3 months 3.Being literate and cooperative 4.Being volunteer 5.Volunteer patients diagnosed with chronic neck pain by a specialist

Inclusion criteria in the control group;

1. Asymptomatic individuals between the ages of 18-64
2. Without any known disease diagnosis and health problems that would affect the evaluations

Exclusion Criteria:

1. Being pregnant,
2. Malignancy,
3. Having cervical stenosis,
4. Severe cervical spondylosis,
5. Cervical fractures and tumor,
6. Osteoporosis,
7. Neurologic deficit related to compression of the spinal root or cord,
8. Having neurologic, dermatologic, infectious, inflammatory rheumatologic and endocrine diseases,
9. Any problems that will hinder exercise (advanced cardiopulmonary or orthopedic problems), having intervention including exercise program or physiotherapy in the three months

Exclusion criteria for the control group; People with cognitive, orthopaedic or neurological diseases that could negatively affect the evaluations

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Between the ages of 18-64 men and women.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Balance | Baseline
  The Biodex Balance System (BBS; Biodex Medical Systems, Shirley, New York, USA) was used to assess postural control.The evaluated parameters of this system are presented below:The modified clinical test of sensory integration of balance (mCTSIB), athletic single leg test (ASLT), limits of stability (LOS), and fall risk assessment were performed with and without a cognitive task.
The modified Clinical Test of Sensory Integration of Balance (mCTSIB) | Baseline
  The mCTSIB was used to assess individuals capability to use sensory inputs for balance.
Athletic Single Leg Test (ASLT) | Baseline
  The evaluation was made with eyes open and closed on one leg (dominant limb) on a firm floor on the balance device platform
Limits of Stability (LOS): | Baseline
  This test is the best test that measures dynamic control among the standard sway tests.
Fall risk assessment | Baseline
  The pre-test platform level was adjusted so that the starting position was 12 and the ending position was 8

SECONDARY OUTCOMES:
Disability level | Baseline
  The disability level will be measured with the Turkish version of Neck Disability Index (NDI). It consists of 10 sections which include the severity of pain, personal care, lifting, reading, headache, concentration, work-life, driving, sleeping and leisure activities. There are 6 responses for each section, scored 0 (no pain and no functional limitation) and 5 (worst pain and maximum limitation). The total score ranges from 0 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet G KARAKAYA, Prof, PT, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Hayriye Yılmaz, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No